CLINICAL TRIAL: NCT01267045
Title: A Randomized Controlled Trial of a Mindfulness Based Intervention for Gulf War Syndrome
Brief Title: Mindfulness-Based Stress Reduction for Gulf War Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPLD-008-10S
Record Dates: First submitted 2010-12-23; First posted 2010-12-24 (Estimated); Results first posted 2014-12-17 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-07

CONDITIONS: Persian Gulf Syndrome
Keywords: Persian Gulf Syndrome; Pain; Fatigue; Attention; Meditation
MeSH Terms: conditions — Persian Gulf Syndrome; Pain; Fatigue | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Participants in this arm undergo the mindfulness training intervention through taking part in a Mindfulness-Based Stress Reduction course
  Interventions: Behavioral: Mindfulness-based stress reduction
- Arm 2 (No Intervention): Treatment as usual for Gulf War Syndrome symptoms (medications, psychotherapy, etc.)

INTERVENTIONS:
Behavioral: Mindfulness-based stress reduction — Mindfulness-Based Stress Reduction (MBSR) teaches mindfulness as a non-religious practice of self-observation and self-awareness. Kabat-Zinn developed MBSR in 1979 in response to a growing awareness that medical interventions were often inadequate at addressing chronic pain issues and restoring function and life satisfaction. He drew on his meditation and yoga training to develop this program as a complement to traditional medicine that could help patients live fully despite their chronic medical and psychiatric conditions. Through MBSR an individual's emphasis shifts from a preoccupation with what is wrong to a growing appreciation for what is right and what can be built upon.
  Arms: Arm 1

SUMMARY:
This pilot study is a two arm randomized, controlled clinical trial that evaluated whether a standardized Mindfulness-Based Stress Reduction (MBSR) intervention reduces symptoms associated with Gulf War Syndrome (GWS) more effectively than treatment as usual. Fifty-five veterans meeting diagnostic criteria for Gulf War Syndrome were randomized to treatment as usual (TAU) or TAU plus an 8-week course of course of MBSR. Study measures were collected at baseline, immediate post-MBSR, and 6 months post intervention. Measures were obtained at equivalent time points for veterans randomized to TAU only. Following completion of all study activities, veterans randomized to TAU only had the opportunity to enroll in MBSR.

DETAILED DESCRIPTION:
A randomized controlled trial with two arms. 55 veterans meeting diagnostic criteria for Gulf War Syndrome were randomized to standard care or standard care plus an 8-week course of course of Mindfulness-Based Stress Reduction (MBSR). Study measures were collected at baseline, immediate post-MBSR (within one week of completion of the MBSR class) and 6 months following completion of the MBSR course. Measures were obtained at equivalent time points for veterans randomized to usual care only. Following completion, veterans randomized to standard care only had the opportunity to enroll in MBSR.

This pilot study will whether there is sufficient evidence of benefit to warrant further study, and gathered data that will allow estimation of the sample size needed in future studies. We also obtained measures working memory and attention, in addition to patient self-report measures of symptoms, in order to provide additional assessment of whether MBSR is effective. This project is prerequisite to a larger study.

ELIGIBILITY:
Inclusion Criteria:

Chart Diagnosis of PTSD

Exclusion Criteria:

* any past or present psychiatric disorder involving a history of psychosis (schizophrenia, schizoaffective disorder, delusional disorder, psychotic disorder not otherwise specified, etc.)
* Mania or poorly controlled bipolar
* Current suicidal or homicidal ideation
* Prior training in mindfulness meditation
* Active substance abuse or dependence
* Must not have had an inpatient admission for psychiatric reasons within the past month

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2010-10; Primary Completion 2012-12 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J Kearney, MD, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Participants in this arm undergo the mindfulness training intervention through taking part in a Mindfulness-Based Stress Reduction.
  Mindfulness-based stress reduction: A common clinical method of teaching mindfulness is a class series called "mindfulness-based stress reduction" (MBSR), which is available at over 250 hospitals nationwide. MBSR teaches mindfulness as a non-religious practice of self-observation and self-awareness. Kabat-Zinn developed MBSR in 1979 in response to a growing awareness that medical interventions were often inadequate at addressing chronic pain issues and restoring function and life satisfaction. He drew on his meditation and yoga training to develop this program as a complement to traditional medicine that could help patients live fully despite their chronic medical and psychiatric conditions. Through MBSR an individual's emphasis shifts from a preoccupation with what is wrong to a growing appreciation for what is right and what can be built upon.
Period: 2-month Outcomes
Arm/Group | Arm 1 | Arm 2
Started | 26 | 29
Completed | 22 | 26
Not Completed | 4 | 3
Period: 6-month Outcome
Arm/Group | Arm 1 | Arm 2
Started | 22 | 26
Completed | 22 | 23
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Participants in this arm undergo the mindfulness training intervention through taking part in Mindfulness-Based Stress Reduction.
  Mindfulness-based stress reduction: A common clinical method of teaching mindfulness is a standardized class called "mindfulness-based stress reduction" (MBSR), which is available at over 250 hospitals nationwide. MBSR teaches mindfulness as a non-religious practice of self-observation and self-awareness. Kabat-Zinn developed MBSR in 1979 in response to a growing awareness that medical interventions were often inadequate at addressing chronic pain issues and restoring function and life satisfaction. He drew on his meditation and yoga training to develop this program as a complement to traditional medicine that could help patients live fully despite their chronic medical and psychiatric conditions. Through MBSR an individual's emphasis shifts from a preoccupation with what is wrong to a growing appreciation for what is right and what can be built upon.
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 26 | 29 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 29 | 54
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (6.8) | 48.6 (7.4) | 49.9 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 23 | 24 | 47
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 8 | 10
  White | 17 | 17 | 34
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 1 | 7
Region of Enrollment [Number; unit: participants]
  United States | 26 | 29 | 55
McGill Pain Questionnaire score [Mean (Standard Deviation); unit: units on a scale] — The Short-Form McGill Pain Questionnaire is a self-report 22-item measure that assesses various types of pain on a scale of 0 (none) to 10 (worst possible) experienced during the past week.
  units on a scale | 75 (32.5) | 81.2 (41.9) | 77.1 (31.3)
Multidimensional Fatigue Inventory [Mean (Standard Deviation); unit: units on a scale] — The Multidimensional Fatigue Inventory is a 20-item self-report measure of various types of fatigue. Each item is a statement, and the subject indicates how much, on a scale of 1 (yes, that is true) to 5 (no, that is not true), he or she agrees with the statement (e.g. "I feel very active.")
  units on a scale
    General Fatigue | 16.0 (2.8) | 15.5 (3.2) | 15.8 (3.0)
    Physical Fatigue | 14.4 (2.7) | 15.3 (2.9) | 14.9 (2.8)
    Reduced Activity | 14.9 (4.1) | 14.3 (3.8) | 14.6 (3.9)
    Reduced Motivation | 11.5 (2.4) | 11.6 (2.4) | 11.5 (2.4)
    Mental Fatigue | 15.5 (3.6) | 15.6 (3.2) | 15.5 (3.3)
Cognitive Failures Questionnaire [Mean (Standard Deviation); unit: units on a scale] — The Cognitive Failure Questionnaire is a 25-item self-report measure of cognitive difficulty during daily living in the past six months. Each item is a question indicating a situation involving a type of cognitive failure (e.g. "Do you find you forget why you went from one part of the house to another?"), and the subject indicates how often that happens to them, on a scale of 0 (never) to 4 (very often).
  units on a scale | 59.6 (16.5) | 58.3 (18.7) | 58.9 (17.5)
PTSD Symptom Scale Interview [Mean (Standard Deviation); unit: units on a scale] | 29 (11.2) | 26.2 (10.6) | 27.5 (10.9)
Medication Use at Baseline [Number; unit: participants] — This is a summary of the prevalence of medication use among the study participants. Since each participant could endorse anywhere from none of these medications to all four types of medication, the total number is unlikely to add up to the exact number of participants.
  participants
    Opiate | 14 | 5 | 19
    Antidepressant | 13 | 14 | 27
    Benzodiazepine | 4 | 4 | 8
    Amphetamine | 2 | 3 | 5
Musculoskeletal Pain [Number; unit: participants]
  Current musculoskeletal pain diagnosis | 20 | 27 | 47
  No musculoskeletal pain diagnosis | 6 | 2 | 8
Neurologic Pain [Number; unit: participants]
  Current neurologic pain diagnosis | 14 | 15 | 29
  No neurologic pain diagnosis | 12 | 14 | 26
Gastrointestinal Condition [Number; unit: participants]
  Current GI condition diagnosis | 10 | 19 | 29
  No GI condition diagnosis | 16 | 10 | 26
Respiratory Conditions [Number; unit: participants]
  Current respiratory condition diagnosis | 10 | 12 | 22
  No respiratory condition diagnosis | 16 | 17 | 33

OUTCOME MEASURES:

1. Primary Outcome: The Short-form McGill Pain Questionnaire
Description: The Short-Form McGill Pain Questionnaire is a self-report 22-item measure that assesses various types of pain on a scale of 0 (none) to 10 (worst possible) experienced during the past week. Score ranges from a minimum of 0 to a maximum of 220; the higher the score, the worse the outcome.
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Arm 1: Participants in this arm undergo the mindfulness training intervention through taking part in a Mindfulness-Based Stress Reduction course
  The most common clinical method of teaching mindfulness is a standardized class called "mindfulness-based stress reduction" (MBSR), which is available at over 250 hospitals nationwide. MBSR teaches mindfulness as a non-religious practice of self-observation and self-awareness. Kabat-Zinn developed MBSR in 1979 in response to a growing awareness that medical interventions were often inadequate at addressing chronic pain issues and restoring function and life satisfaction. He drew on his meditation and yoga training to develop this program as a complement to traditional medicine that could help patients live fully despite their chronic medical and psychiatric conditions. Through MBSR an individual's emphasis shifts from a preoccupation with what is wrong to a growing appreciation for what is right and what can be built upon.
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 22 | 26
units on a scale | 54.0 (44.2) | 65.5 (43.4)

2. Secondary Outcome: Patient Health Questionnaire (PHQ-9)
Description: The Patient Health Questionnaire (PHQ-9) is a 9-item (with an additional 10th item if any of the previous 9 are endorsed) self-report measure of depression. Subjects are instructed to indicate how often, over the last 2 weeks, they have been bothered by each problem (e.g. "feeling tired or having little energy"), from "not at all" (0), to "nearly every day" (3). Scores range from a minimum of 0 to a maximum of 30; the higher the score, the worse the outcome.
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Arm 1: Participants in this arm undergo the mindfulness training intervention through taking part in a Mindfulness-Based Stress Reduction course
  The most common clinical method of teaching mindfulness is a standardized class called "mindfulness-based stress reduction" (MBSR), which is available at over 250 hospitals nationwide. MBSR teaches mindfulness as a non-religious practice of self-observation and self-awareness. Kabat-Zinn developed MBSR in 1979 in response to a growing awareness that medical interventions were often inadequate at addressing chronic pain issues and restoring function and life satisfaction. He drew on his meditation and yoga training to develop this program as a complement to traditional medicine that could help patients live fully despite their chronic medical and psychiatric conditions. Through MBSR an individual's emphasis shifts from a preoccupation with what is wrong to a growing appreciation for what is right and what can b
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 22 | 26
units on a scale | 10.2 (6.2) | 12.4 (6.7)

3. Primary Outcome: The Short-Form McGill Pain Questionnaire
Description: as for outcome 1
Time Frame: 8 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 22 | 23
units on a scale | 57.1 (44.7) | 76.6 (49.3)

4. Primary Outcome: Multidimensional Fatigue Inventory - General Fatigue
Description: The Multidimensional Fatigue Inventory is a 20-item self-report measure of various types of fatigue. Each item is a statement, and the subject indicates how much, on a scale of 1 (yes, that is true) to 5 (no, that is not true), he or she agrees with the statement (e.g. "I feel very active.") Scores range from a minimum of 20 to a maximum of 100; the higher the score, the worse the outcome.
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 22 | 26
units on a scale | 14.9 (3.6) | 15.5 (2.9)

5. Primary Outcome: Multidimensional Fatigue Inventory - General Fatigue
Description: as for outcome 4
Time Frame: 8 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 22 | 23
units on a scale | 13.6 (3.4) | 15.3 (3.6)

6. Primary Outcome: Cognitive Failures Questionnaire
Description: The Cognitive Failure Questionnaire is a 25-item self-report measure of cognitive difficulty during daily living in the past six months. Each item is a question indicating a situation involving a type of cognitive failure (e.g. "Do you find you forget why you went from one part of the house to another?"), and the subject indicates how often that happens to them, on a scale of 0 (never) to 4 (very often). Scores range from a minimum of 0 to a maximum of 100; the higher the score, the worse the outcome.
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 22 | 26
units on a scale | 46.9 (18.1) | 58.6 (18.1)

7. Primary Outcome: Cognitive Failures Questionnaire
Description: as for outcome 6
Time Frame: 8 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 22 | 23
units on a scale | 46.6 (15.4) | 61.9 (18.6)

8. Secondary Outcome: Patient Health Questionnaire (PHQ-9)
Description: as for outcome 2
Time Frame: 8 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 22 | 23
units on a scale | 9.5 (4.7) | 12.3 (6.8)

9. Secondary Outcome: PTSD Symptom Severity Interview (PSSI)
Description: The PTSD Symptom Severity Interview (PSSI) is a 17-question interview that measures the severity of PTSD symptoms in the past month. The interviewing researcher asks the subject to respond to each question (e.g. "Have you had recurrent or intrusive distressing thoughts or recollections about the trauma?") by indicating how often per week he or she experiences that symptom. For each item, "not at all" is scored as 0; "once per week or less/a little" is scored as 1; "2 to 4 times per week/somewhat" is scored as 2; and "5 or more times per week/very much" is scored as 3. Total scores range from a minimum of 17 to a maximum of 51; the higher the score, the worse the outcome.
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 22 | 26
units on a scale | 20.7 (9.1) | 24.7 (10.2)

10. Secondary Outcome: PTSD Symptom Severity Interview (PSSI)
Description: as for outcome 9
Time Frame: 8 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 22 | 23
units on a scale | 21.7 (10.8) | 23.6 (10.7)

11. Secondary Outcome: PROMIS Fatigue
Description: The self-report PROMIS Fatigue measure uses a maximum of 7 questions to assess fatigue symptoms over the past 7 days. Subjects respond to each question (e.g. "How often did you feel tired?) with the following scale:
  1. = never
  2. = rarely
  3. = sometimes
  4. = often
  5. = always
  Raw scores are converted to T-scores, which are standardized to a mean of 50. Scores above 50 indicate higher than average fatigue; scores below 50 indicate lower than average fatigue.
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 22 | 26
T-score | 56.0 (8.6) | 61.5 (9.3)

12. Secondary Outcome: PROMIS Fatigue
Description: as for outcome 11
Time Frame: 8 months
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 22 | 23
T-score | 57.5 (9.6) | 62.0 (10.0)

13. Secondary Outcome: Five Facet Mindfulness Questionnaire
Description: The Five Facet Mindfulness Questionnaire (FFMQ) measures five aspects of mindfulness: Observing, Describing, Acting with Awareness, Non-judging, and Non-reacting. It is a 39-item self-report questionnaire. Subjects respond to each statement (e.g. "I disapprove of myself when I have irrational ideas") by indicating how often they agree with the statement on a scale of 1 ("never or very rarely true") to 5 ("very often or always true"). Scores range from a minimum of 39 to a maximum of 195. Higher scores indicate greater levels of mindfulness.
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 22 | 26
units on a scale | 126.5 (22.7) | 115.0 (15.1)

14. Secondary Outcome: Five Facet Mindfulness Questionnaire
Description: as for outcome 13
Time Frame: 8 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 22 | 23
units on a scale | 129.4 (22.4) | 114.6 (19.6)

ADVERSE EVENTS:
Groups:
- Arm 1: Participants in this arm undergo the mindfulness training intervention through taking part in a Mindfulness-Based Stress Reduction course.
  The most common clinical method of teaching mindfulness is a standardized class called "mindfulness-based stress reduction" (MBSR), which is available at over 250 hospitals nationwide. MBSR teaches mindfulness as a non-religious practice of self-observation and self-awareness. Kabat-Zinn developed MBSR in 1979 in response to a growing awareness that medical interventions were often inadequate at addressing chronic pain issues and restoring function and life satisfaction. He drew on his meditation and yoga training to develop this program as a complement to traditional medicine that could help patients live fully despite their chronic medical and psychiatric conditions. Through MBSR an individual's emphasis shifts from a preoccupation with what is wrong to a growing appreciation for what is right and what can b
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 0/26 | 2/29
Other Adverse Events (participants affected / at risk) | 0/26 | 0/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=26) | Arm 2 (N=29)
Chest pains (Cardiac disorders) | 0 (0) | 1 (1) — The patient was admitted to Tacoma General Hospital for chest pain. He is reported to have had a small cardiac event, and had sent placed as treatment. The IRB determined that this event was probably NOT related to the study.
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) — A participant expressed having suicidal and homicidal ideation during a follow-up assessment. The interview was terminated and the researcher escorted the patient to psychiatric emergency services.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes